CLINICAL TRIAL: NCT01303029
Title: A Phase IIb Randomized Study to Evaluate the Efficacy of Gemcitabine-erlotinib Versus Gemcitabine-erlotinib-capecitabine in Patients With Metastatic Pancreatic Cancer
Brief Title: Safety and Efficacy Study of Gemcitabine-erlotinib Versus Gemcitabine-erlotinib-capecitabine in Patients With Metastatic Pancreatic Cancer
Acronym: GECA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTD-10-01; 2010-022599-30 (EudraCT Number)
Record Dates: First submitted 2011-02-16; First posted 2011-02-24 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Pancreatic cancer; gemcitabine; erlotinib; capecitabine
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Gemcitabine+erlotinib
  Interventions: Drug: Gemcitabine+erlotinib
- Experimental (Experimental): Gemcitabine+erlotinib+capecitabine
  Interventions: Drug: Gemcitabine+erlotinib+capecitabine

INTERVENTIONS:
Drug: Gemcitabine+erlotinib — Gemcitabine 1000mg/m2 over 30 minutes on days 1, 8, 15. Erlotinib will be administered orally at a dose of 100 mg daily from day 1 to day 28, repeated every 4 weeks .
  Arms: Control
Drug: Gemcitabine+erlotinib+capecitabine — Gemcitabine 1000mg/m2 over 30 minutes on days 1, 8, 15. Capecitabine will be administered orally 1.660 mg/m2 day from day 1 to day 21. Erlotinib will be administered orally at a dose of 100 mg daily from day 1 to day 28, repeated every 4 weeks .
  Arms: Experimental

SUMMARY:
The purpose of the study is to evaluate the efficacy of the combination of gemcitabine-erlotinib versus gemcitabine-erlotinib-capecitabine in patients with metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent
2. Able, in the investigator's opinion, to fulfill the procedures and explorations of the study
3. Age ≥ 18 years old
4. ECOG 0-2
5. Life expectancy ≥ 12 weeks
6. Patients with metastatic adenocarcinoma of the pancreas, following 7th edition of TNM classification
7. Histologically or cytologically confirmed diagnosis of adenocarcinoma of the pancreas
8. Measurable disease following RECIST criteria version 1.1
9. No previous systemic treatment for metastatic pancreatic cancer Adjuvant chemotherapy al least 6 months before enrollment is allowed. Patients having neoadjuvant chemotherapy must have completed the treatment at least 4 weeks before trial entry. Toxicities associated to previous treatment must be resolved before enrollment. Progression disease (metastatic disease) must be confirmed after adjuvant treatment
10. Adequate bone marrow function as determined by:

    * Hemoglobin: ≥ 9 g/dL. (patients with hemoglobin < 9 g/dL could be transfused before their inclusion on the study)
    * Platelets: ≥ 100 x 109/L
    * Absolute Neutrophil account (ANC) ≥ 1,5 x 109/L
11. Adequate liver function, as determined by:

    * Serum bilirubin ≤ 1,5 x LSN
    * AST, ALT ≤ 2,5 x LSN in patients without liver metastasis. In patients with liver metastasis ≤ 5 x LSN
    * Alkaline phosphatase ≤ 2,5 x LSN or ≤ 5 x LSN in patients with liver metastasis. In patients with bone metastasis ≤ 10 x LSN
12. Adequate renal function, as determined by:

    * Creatinine clearance using the Cockcroft-Gault formula ≥ 50.0 ml/min
13. Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to randomization. Postmenopausal women are defined as those who have been amenorrheic for at least 12 months. Also, both men and women enrolled in this study must use adequate birth control (eg., abstinence, intrauterine device, oral contraceptive or double barrier method or be surgically sterile), starting at the signing of the informed consent and up to at least 6 months after completion of treatment or the last dose, whichever occurs first
14. Patients must not have undergone a major surgical procedure within 4 weeks prior to study treatment. The surgical wound should be completely healed

Exclusion Criteria:

1. Local pancreatic cancer (stage IA-IIB) or locally advance cancer (stage III), following the TNM 7th edition classification. Patients with metastatic disease that relapse after the initial diagnosis of local or advance disease could be included in this study
2. Pancreatic endocrine tumor and ampulloma
3. Evidence of carcinomatosis meningitis or brain metastasis. In case of clinical suspicious of brain metastasis is mandatory to perform a brain TAC/MR 4 weeks prior de inclusion.
4. Primary tumors developed 5 years previous to the inclusion, except in situ cervix carcinoma or skin basocellular cancer properly treated
5. Cardiovascular disease clinically significant (active):

   * Non-controlled arterial hypertension (Systolic pressure > 150 mg Hg and/or diastolic pressure > 100 mm Hg on repeated pressure measurements)
   * Cerebrovascular accident/ictus (≤ 6 weeks prior to inclusion)
   * Myocardial infarction (≤ 6 months prior to inclusion)
   * Unstable angina
   * Congestive cardiac insufficiency (grade II or superior following to New York Heart Association (NYHA)
   * Severe cardiac arrythmia requiring treatment
6. Significant ophthalmologic anomalies
7. Deficit in Dihydropyrimidine-Dehydrogenase (DPD)
8. Unable to take oral drug. Previous surgical process that affect the absorption or make the needed to have intravenous feeding or parenteral nutrition with lipids
9. Pregnancy women or in lactation period
10. Antineoplastic treatment (chemotherapy, hormonal treatment, radiotherapy, surgery, biological therapy or tumor embolization) 4 weeks prior the inclusion
11. Previous treatment with capecitabine or EGFR inhibitor
12. Metabolic disease or any other disease which, in the investigator's opinion, might interfere with the treatment in study
13. Known hypersensibility to any study drug (gemcitabine, erlotinib, capecitabine) or to 5-fluorouracile and fluoropyrimidines
14. Current infection grade ≥ 2 (CTCAE)
15. Known human immunodeficiency virus infection, or chronic infection with hepatitis B or C virus, or severe uncontrolled intercurrent infection or other severe uncontrolled concomitant diseases
16. Medical, psychological, psychiatric or sociological conditions that would interfere to the patient participation in the study or in the assessment of the results
17. Current or 30 days previous to study treatment with other investigational drug or participation in other trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 4 years

SECONDARY OUTCOMES:
Overall survival | 4 years
Response rate (RR) | 4 years
Duration of response | 4 years
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 4 years
Percentage of rash in patients treated with erlotinib and progression free survival and overall survival and treatment relationship | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Irigoyen, MD, Study Chair — Hospital de Toledo, Spain; Manuel Benavides, MD, Study Chair — Hospital Carlos Haya, Málaga. Spain
Locations (1):
- Spanish Cooperative Group for Digestive Tumour Therapy, Madrid, Spain

REFERENCES:
- [Derived] Irigoyen A, Gallego J, Guillen Ponce C, Vera R, Iranzo V, Ales I, Arevalo S, Pisa A, Martin M, Salud A, Falco E, Saenz A, Manzano Mozo JL, Pulido G, Martinez Galan J, Pazo-Cid R, Rivera F, Garcia Garcia T, Serra O, Fernandez Parra EM, Hurtado A, Gomez Reina MJ, Lopez Gomez LJ, Martinez Ortega E, Benavides M, Aranda E; Spanish Cooperative Group of Treatment of Digestive Tumors (TTD). Gemcitabine-erlotinib versus gemcitabine-erlotinib-capecitabine in the first-line treatment of patients with metastatic pancreatic cancer: Efficacy and safety results of a phase IIb randomised study from the Spanish TTD Collaborative Group. Eur J Cancer. 2017 Apr;75:73-82. doi: 10.1016/j.ejca.2016.12.032. Epub 2017 Mar 7. PMID 28222309
- See also: Related Info — http://www.ttdgroup.org